CLINICAL TRIAL: NCT02039336
Title: Phase I/II Study With the Combination of Dacomitinib and PD-0325901 in Metastatic KRAS Mutation Positive Non-small Cell Lung Cancer
Brief Title: Dacomitinib Plus PD-0325901 in Advanced KRAS Mutant NSCLC
Acronym: M13DAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL45985.031.13
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — dacomitinib; mirdametinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dacomitinib + PD-0325901 (Experimental): Dacomitinib: oral tablets PD-0325901: oral capsules
  Interventions: Drug: Dacomitinib; Drug: PD-0325901; Drug: Docetaxel

INTERVENTIONS:
Drug: Dacomitinib
Drug: PD-0325901
Drug: Docetaxel

SUMMARY:
This is a phase I/II multi-center open-label proof of concept study, consisting of two parts. Part A of this study is designed to identify the recommended phase 2 dose (RP2D) of the combination regimen of dacomitinib plus PD-0325901 in patients with advanced KRAS mutant (KRASm) non-small cell lung cancer (NSCLC). Part B is designed to perform a randomized comparison of the combination of dacomitinib and PD-0325901 versus standard of care therapy in patients with advanced KRASm NSCLC. It is hypothesized that with this combination strategy the progression free survival of patients with KRASm NSCLC will be doubled.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of advanced non-small cell lung cancer
* Written documentation of KRAS (exon 2, 3 or 4) mutation
* At least 18 years of age or older
* Able and willing to give written informed consent
* WHO performance status of 0 or 1

Exclusion Criteria:

* Symptomatic or untreated leptomeningeal disease
* Symptomatic brain metastasis
* Impairment of gastrointestinal function
* Uncontrolled infectious disease
* Left ventricular ejection fraction < 50%
* Retinal degenerative disease or with history of uveitis, retinal vein occlusion or retinal detachment

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose-limiting toxicities | 1.5 years
Progression free survival | 2.5 years

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 2.5 years
Plasma concentration | 2.5 years
Overall response rate | 2.5 years
Duration of response | 1.5 years
Time to response | 2.5 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: f opdam, MD, PhD, Study Director — The Netherlands Cancer Institute; FALM Eskens, PhD, Principal Investigator — Erasmus Medical Centre Cancer Institute; MPJK Lolkema, PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Netherlands (3):
  - The Netherlands Cancer Institute, Amsterdam
  - Erasmus Medical Center Cancer Institute, Rotterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] van Geel RMJM, van Brummelen EMJ, Eskens FALM, Huijberts SCFA, de Vos FYFL, Lolkema MPJK, Devriese LA, Opdam FL, Marchetti S, Steeghs N, Monkhorst K, Thijssen B, Rosing H, Huitema ADR, Beijnen JH, Bernards R, Schellens JHM. Phase 1 study of the pan-HER inhibitor dacomitinib plus the MEK1/2 inhibitor PD-0325901 in patients with KRAS-mutation-positive colorectal, non-small-cell lung and pancreatic cancer. Br J Cancer. 2020 Apr;122(8):1166-1174. doi: 10.1038/s41416-020-0776-z. Epub 2020 Mar 9. PMID 32147669